CLINICAL TRIAL: NCT01701505
Title: A Phase 2, Single-Center, Open-Label, Randomized, Parallel-Groups, Dose-Ranging Study to Assess the Efficacy and Safety of Intranasally Administered Kovacaine Mist for Anesthetizing Maxillary Teeth in Pediatric Subjects
Brief Title: Dose-Ranging Study of Intranasal Kovacaine Mist in Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR 2-03
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
Keywords: operative; dental procedure
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kovacaine Mist High Dose (Experimental): 400uL of Kovacaine Mist, as 2 sprays of 200uL.
  Interventions: Drug: 400uL of Kovacaine Mist
- Kovacaine Mist Mid Dose (Experimental): 200uL of Kovacaine Mist, as 2 sprays of 100uL.
  Interventions: Drug: 200uL of Kovacaine Mist
- Kovacaine Mist Low Dose (Experimental): 120uL of Kovacaine Mist, as 2 sprays of 60uL.
  Interventions: Drug: 120uL of Kovacaine Mist

INTERVENTIONS:
Drug: 400uL of Kovacaine Mist — 2 unilateral intranasal sprays of 200uL each.
  Other Names: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
  Arms: Kovacaine Mist High Dose
Drug: 200uL of Kovacaine Mist — 2 unilateral intranasal sprays of 100uL each.
  Other Names: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
  Arms: Kovacaine Mist Mid Dose
Drug: 120uL of Kovacaine Mist — 2 unilateral intranasal sprays of 60uL each.
  Other Names: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
  Arms: Kovacaine Mist Low Dose

SUMMARY:
The purpose of this study is to assess the efficacy and safety of intranasally administered Kovacaine Mist for anesthetizing maxillary teeth in pediatric subjects.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, parallel-groups, dose-ranging study to assess the efficacy and safety of intranasally administered Kovacaine Mist for anesthetizing maxillary teeth in pediatric subjects.

The study will employ an open-label design to determine the lowest effective doses (LEDs), and assess the safety and efficacy of Kovacaine Mist administered intranasally for inducing pulpal anesthesia of maxillary primary teeth numbers A to J and maxillary permanent teeth numbers 4 to 13 (maxillary right second premolar to maxillary left second premolar) sufficient to allow completion of the Study Dental Procedure, and will be carried out in healthy children of either sex between the ages of 3 and 17 years, inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 3-17 years of age inclusive.
* Need for an operative restorative dental procedure on a single vital maxillary primary tooth (#A to J) or permanent tooth (#4 to13), other than a maxillary permanent first, second or third molar, requiring local anesthesia with an expected treatment duration not exceeding 60 minutes.
* Normal lip, nose, eyelid, and cheek sensation.
* Accompanied and/or represented by a parent or guardian able to comprehend and sign the informed consent document.
* If age 8 and above, able to understand and provide informed assent.
* Patient or parent/guardian able to communicate with the investigator and comply with the requirements of the protocol.
* Patency of the naris ipsilateral to the tooth undergoing the Study Dental Procedure.
* Minimum weight: Subjects in Cohorts A and B (age 6 and above) must weigh at least 20kg (44 lb.). Subjects in Cohort C (age 3 and above) must weigh at least 10kg (22 lb.).

Exclusion Criteria:

* Dental care requiring a local anesthetic within the 24 hours prior to anticipated study participation.
* History of allergy to or intolerance of tetracaine, benzyl alcohol, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreen).
* History of allergy or hypersensitivity to lidocaine, oxymetazoline, epinephrine, or sulfite preservatives.
* Use of a monoamine oxidase inhibitor within the 3 weeks preceding study entry.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females of child-bearing potential will be required to take a urine pregnancy test on the day of, but prior to, study drug administration to rule out pregnancy.)
* Inadequately controlled thyroid disease of any type.
* Use of any investigational drug (including Kovacaine Mist) and/or participation in any clinical trial within 30 days of study participation.
* Frequent nose bleeds (≥ 5 per month).
* Anticipated need for use of oxymetazoline or phenylephrine nasal spray, nasal irrigation, or other nasal or oral decongestant on the day of the study procedure.
* History of congenital or idiopathic methemoglobinemia.
* Clinically relevant history of sinus/nasal surgery, recent epistaxis, nasal congestion or sinus infections, or use of a "sinus medication" within the 48 hours prior to anticipated study participation.
* History of alcoholism and/or drug abuse.
* Pulpal pathology in the index tooth.
* Anticipated need for use of nitrous oxide before or during the Study Dental Procedure.
* Any chronic or currently uncontrolled psychogenic, neurological, endocrine, pulmonary, cardiovascular, renal, gastrointestinal or hepatic disease or condition with manifestations that might confound interpretation of study results or make receipt of study medication a source of risk for adverse outcome.
* Fever defined as body temperature ≥100° (37°C) on the day of and prior to study drug administration.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Moore, DMD/PhD/MPH, Study Director — University of Pittsburgh
Locations (1):
- Big Grins, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist); Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist): 120uL of Kovacaine Mist: 2 unilateral intranasal sprays of 60uL each.
- Cohort A: 12-17 Years Mid-Dose (200uL Kovacaine Mist); Cohort B: 7-11 Years Med Dose: 200uL of Kovacaine Mist: 2 unilateral intranasal sprays of 100uL each.
- Cohort A: 12-17 Years HighDose (400uL Kovacaine Mist): 400uL of Kovacaine Mist: 2 unilateral intranasal sprays of 200uL each.
- Cohort C: 3-6 Years Low Dose: 120uL of Kovacaine Mist, as 2 sprays of 60uL
  120uL of Kovacaine Mist: 2 unilateral intranasal sprays of 60uL each
Period: Overall Study
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Mid-Dose (200uL Kovacaine Mist) | Cohort A: 12-17 Years HighDose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose | Cohort C: 3-6 Years Low Dose
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist); Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist): 200uL of Kovacaine Mist: 2 unilateral intranasal sprays of 100uL each
- Cohort A: 12-17 High Dose (400uL Kovacaine Mist): 400uL of Kovacaine Mist: 2 unilateral intranasal sprays of 200uL each
- Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist): 120uL of Kovacaine Mist: 2 unilateral intranasal sprays of 60uL each
- Total: Total of all reporting groups
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.75) | 14.4 (2.00) | 13.6 (1.19) | 8.9 (1.64) | 7.9 (0.83) | 5.3 (1.04) | 10.7 (3.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 3 | 6 | 5 | 2 | 28
  Male | 4 | 0 | 5 | 2 | 3 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 2 | 0 | 1 | 9
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 8 | 7 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 5 | 7 | 6 | 8 | 7 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 2 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic.
Description: If the participant does not have sufficient anesthesia to complete the Study Dental Procedure, the participant is given a rescue injection of local anesthetic and is considered a failure for this outcome.
Time Frame: at 14 minutes with a 3 minute window
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants | 6 | 7 | 8 | 5 | 7 | 4

2. Secondary Outcome: Naris Examination (NE) to Assess Reactions to the Study Drug.
Description: The principal investigator will perform a visual inspection to note number of participants at post-dose that have a ulceration, inflammation or minor bleeding.
Time Frame: At Baseline and 120 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants
  Post-dose ulceration (not present at baseline | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose inflammation (not present at baseli | 0 | 1 | 0 | 0 | 0 | 0
  Post-dose minor bleeding (not present at baseline) | 1 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Systolic Blood Pressure
Time Frame: At Baseline, 12 minutes, and 120 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
mmHg
  Baseline | 113.1 (8.44) | 122.5 (11.41) | 115.4 (10.06) | 111.3 (7.59) | 106.5 (9.35) | 97.8 (8.36)
  12 mins | 119.1 (12.19) | 122.3 (10.89) | 121.0 (21.21) | 105.5 (13.32) | 109.9 (6.53) | 101.9 (10.19)
  120 mins | 120.5 (9.27) | 120.1 (10.32) | 116.4 (9.62) | 106.3 (8.84) | 102.3 (9.81) | 101.9 (16.16)

4. Secondary Outcome: Diastolic Blood Pressure
Time Frame: At Baseline, 12 minutes, and 120 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
mmHg
  Baseline | 64.6 (6.93) | 70.9 (7.16) | 62.1 (9.37) | 65.0 (11.71) | 63.8 (6.96) | 61.0 (8.19)
  12 mins | 63.9 (3.40) | 68.4 (7.85) | 66.1 (10.96) | 62.0 (6.78) | 64.6 (4.78) | 60.4 (7.93)
  120 mins | 64.3 (10.67) | 69.0 (10.57) | 70.1 (8.51) | 65.0 (6.41) | 61.6 (8.47) | 66.1 (13.58)

5. Secondary Outcome: Heart Rate
Time Frame: At Baseline, 12 minutes, and 120 minutes
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
bpm
  Baseline | 72.9 (10.55) | 83.6 (12.95) | 75.5 (14.80) | 90.3 (15.04) | 80.6 (7.41) | 90.1 (7.66)
  12 mins | 75.4 (10.06) | 80.9 (12.43) | 77.3 (18.52) | 91.6 (15.14) | 82.5 (9.01) | 89.3 (11.59)
  120 mins | 78.4 (11.02) | 84.3 (14.58) | 76.1 (10.45) | 91.9 (13.01) | 86.9 (7.10) | 95.0 (4.54)

6. Secondary Outcome: Oxygen Saturation
Time Frame: At Baseline, 12 minutes, and 120 minutes
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percent
  Baseline | 97.3 (1.28) | 98.8 (1.75) | 98.3 (1.39) | 97.3 (1.49) | 97.4 (2.00) | 97.6 (1.30)
  12 mins | 97.3 (1.28) | 98.3 (1.49) | 97.9 (1.36) | 97.4 (1.30) | 96.3 (2.19) | 96.4 (0.74)
  120 mins | 97.0 (0.93) | 97.4 (1.51) | 96.9 (1.64) | 96.0 (1.85) | 97.5 (1.31) | 97.5 (1.41)

7. Secondary Outcome: Number of Participants With Adverse Events by Dose Level and Age
Time Frame: from baseline to 24 hours following drug administration
Population: Patients grouped by age
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist High Dose | Kovacaine Mist Mid Dose | Kovacaine Mist Low Dose
Number analyzed (Participants) | 8 | 16 | 24
Participants
  3-6 Years: number analyzed (Participants) | 0 | 0 | 8
  3-6 Years |  |  | 8
  7-11 Years: number analyzed (Participants) | 0 | 8 | 8
  7-11 Years |  | 7 | 6
  12-17 Years: number analyzed (Participants) | 8 | 8 | 8
  12-17 Years | 8 | 5 | 6

8. Secondary Outcome: Incidence of Adverse Events by Dose Level Regardless of Age
Time Frame: from baseline to 24 hours following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist High Dose | Kovacaine Mist Mid Dose | Kovacaine Mist Low Dose
Number analyzed (Participants) | 8 | 16 | 24
Participants | 8 | 12 | 20

ADVERSE EVENTS:
Time Frame: 24 hours post-dosing
Arm/Group | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 5/8 | 8/8 | 6/8 | 7/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: 12-17 Years Low Dose (120uL Kovacaine Mist) (N=8) | Cohort A: 12-17 Years Med Dose (200 uL Kovacaine Mist) (N=8) | Cohort A: 12-17 High Dose (400uL Kovacaine Mist) (N=8) | Cohort B: 7-11 Years Low Dose (120uL Kovacaine Mist) (N=8) | Cohort B: 7-11 Years Med Dose (200 uL Kovacaine Mist) (N=8) | Cohort C: 3-6 Years Low Dose (120uL Kovacaine Mist) (N=8)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 5 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1 | 2 | 2
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 1
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation Increased (Eye disorders) | 1 | 2 | 3 | 5 | 5 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Facial Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intranasal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No